CLINICAL TRIAL: NCT06227091
Title: Analysis of Electromyography Activation Trunk Muscles and the Effect of Beetroot Juice Intake on the Results in Strength Exercises: Lateral Medicine Ball Throw and Sled Pushing
Brief Title: The Effect od Beetroot Juice on Forearm Muscle Strength and Muscle EMG Activity After BloodFlow Restriction
Acronym: BFR_EMG
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Robert Olek, Principal Investigator, Poznan University of Physical Education
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: RMPN2021/JJ2
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Muscle Strength

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot juice (Experimental): beetroot juice with high concentration of nitrates ( 800mg)
  Interventions: Dietary Supplement: Beetroot juice
- Depleted beetroot Juice (Placebo Comparator): beetroot juice with low concentration of nitrates
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beetroot juice — acute dose of beetroot juice
  Arms: Beetroot juice
Dietary Supplement: Placebo — depleted nitrate beetroot juice
  Arms: Depleted beetroot Juice

SUMMARY:
The primary aim of the current study is determine the effect of beetroot juice consumption on maximal grip strength and EMG muscle activity

DETAILED DESCRIPTION:
In random order subjects will consume high nitrate beetroot juice or low level of nitrate beetroot juice. Grip strength and EMG will be measured at the beginning and repeated after 2h.

Using blood pressure cuff, occlusion will be induced to restrict blood flow in the brachial artery. Following the deflation of the cuff, assessments will be conducted for grip strength and electromyography (EMG) activation of the forearm muscles. These measurements will be taken both initially and after a 2-hour interval.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2027-10-20 (Estimated)

PRIMARY OUTCOMES:
The effect of Beetroot Juice consumption on Grip Strength | 2 hours
  Determination of muscle strength following beetroot juice consumption using hand grip dynamometer

SECONDARY OUTCOMES:
The effect of Beetroot Juice consumption on EMG muscle activity | 2 hours
  Determination of forearm muscle activity following beetroot juice consumption using electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Robert Olek, Prof, Principal Investigator — Poznan University of Physical Education
Locations (1):
- Akademia Wychowania Fizycznego, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No